CLINICAL TRIAL: NCT04581824
Title: A Randomized, Phase 2, Double-blind Study to Evaluate the Efficacy of Dostarlimab Plus Chemotherapy Versus Pembrolizumab Plus Chemotherapy in Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Efficacy Comparison of Dostarlimab Plus Chemotherapy Versus Pembrolizumab Plus Chemotherapy in Participants With Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated by GSK for strategic reasons, after all participants completed treatment. This decision was not based on a safety concern
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213403
Record Dates: First submitted 2020-08-31; First posted 2020-10-09 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Non small cell lung cancer; Dostarlimab; Pembrolizumab; Pemetrexed; Carboplatin; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dostarlimab; pembrolizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and study staff may only be blinded to study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving dostarlimab plus chemotherapy (Experimental): Participants will receive dostarlimab on Day 1 of every 21 Day cycle followed by pemetrexed, and then followed by cisplatin or carboplatin (Cycles 1 to 4 only) as per investigator decision.
  Interventions: Drug: Dostarlimab; Drug: Chemotherapy
- Participants receiving pembrolizumab plus chemotherapy (Active Comparator): Participants will receive pembrolizumab on Day 1 of every 21 Day cycle followed by pemetrexed, and then followed by cisplatin or carboplatin (Cycles 1 to 4 only) as per investigator decision.
  Interventions: Drug: Pembrolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab will be administered through a 30 minute infusion at a dose of 500 milligrams (mg) intravenously (IV) every 3 weeks (Q3W) up to a maximum of 35 cycles (each cycle of 21 days).
  Arms: Participants receiving dostarlimab plus chemotherapy
Drug: Pembrolizumab — Pembrolizumab will be administered through a 30 minute infusion at a dose of 200 mg Q3W up to a maximum of 35 cycles (each cycle of 21 days).
  Arms: Participants receiving pembrolizumab plus chemotherapy
Drug: Chemotherapy — Pemetrexed will be administered at 500 milligram per meter square (mg/m^2 ) IV through a 10 minute IV infusion Q3W, up to a maximum of 35 cycles (each cycle of 21 days).
  Cisplatin will be administered at 75 mg/m^2 through a 30 minute IV infusion Q3W for 4 cycles (each cycle of 21 days) as per investigator decision.
  Carboplatin will also be administered at area under the concentration time curve 5 milligram/milliliters/minute (mg/mL/min) (maximum dose: 750 mg) through a 15 to 60 minute IV infusion Q3W for 4 cycles (each cycle of 21 days) as per investigator decision.

SUMMARY:
NSCLC comprises of approximately 84 percent (%) of all lung cancers and is often diagnosed at advanced stage due to poor prognosis. Dostarlimab is an immunoglobulin G (IgG)4 kappa humanized monoclonal antibody (mAb) that binds with high affinity to programmed cell death protein 1 (PD 1), resulting in inhibition of binding to programmed death ligand 1 (PD L1) and programmed death ligand 2 (PD L2). This study aims to compare the efficacy and safety PD-1 inhibitors dostarlimab and pembrolizumab, when administered in combination with chemotherapy (pemetrexed, cisplatin and carboplatin), in participants with non-squamous NSCLC without a known sensitizing epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or receptor tyrosine kinase-1 (ROS-1) mutation, BRAF V600E mutation, or other genomic aberration for which an approved targeted therapy is available. A total of approximately 240 participants will be enrolled in the study for a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than equal to (>=) 18 years old, must be able to understand the study procedures, and agrees to participate in the study by providing written informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participant has histologically- or cytologically-confirmed metastatic non-squamous NSCLC with documented absence of a sensitizing EGFR, ALK, ROS-1, or BRAFV600E mutation or other genomic aberration for which an approved targeted therapy is available. Mixed tumors will be categorized by the predominant cell type; if the tumor has predominantly squamous cell histology or if small cell elements are present, the participant is ineligible.
* Participants must have measurable disease, that is (i.e.) presenting with at least 1 measurable lesion per RECIST v1.1 as determined by the local site Investigator/radiology assessment. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions and if there are other target lesions. If there is only 1 target lesion that was previously irradiated, the participant is not eligible.
* Participant has documented PD L1 status by the 22C3 pharmDx assay (Agilent/Dako). If no prior PD L1 result is available at the time of Screening, the participant can be tested locally using the stated method, or central PD L1 testing can be completed. Results are needed for stratification and must be available prior to randomization.
* Participant has an ECOG performance status score of 0 or 1.
* Participant has a life expectancy of at least 3 months.
* Participant has adequate organ function.
* Participant has recovered to Grade less than equal to (<=)1 from any prior treatment related toxicities at the time of randomization. A participant with Grade 2 alopecia is an exception to this criterion and may qualify for this study.
* Contraceptive use by male and female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants are eligible to participate if they agree to the following during the Treatment Period and for at least 150 days after the last dose of study treatment:
* Refrain from donating sperm plus, either:
* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.
* Must agree to use contraception/barrier as follows:
* Agree to use a male condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception, as a condom may break or leak) when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.
* Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and 1 of the following conditions applies:
* Is a woman of non childbearing potential (WONCBP),
* Is a WOCBP, using a contraceptive method that is highly effective (with a failure rate of <1% per year and, preferably, with low user dependency) during the Treatment Period and for at least 180 days after the last dose of study treatment and agrees not to donate eggs (ova or oocytes) for the purpose of reproduction during this period. The Investigator should evaluate the potential for contraceptive method failure ( for example [e.g.], noncompliance and recently initiated) in relationship to the first dose of study treatment.
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum, as required by local guidelines) within 72 hours before the first dose of study treatment. If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

Exclusion Criteria:

* Participant has received prior systemic therapy for the treatment of metastatic NSCLC. Participants who have received neoadjuvant or adjuvant chemotherapy are eligible if the neoadjuvant/adjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
* Participant has received prior therapy with a PD (L)1 or PD L2 inhibitor, a cytotoxic T lymphocyte associated protein 4 (CTLA 4) inhibitor, a T cell immunoglobulin and mucin domain containing 3 (TIM 3) inhibitor, or any other immunotherapy agent (eg, OX40) for the treatment of cancer.
* Participant has received radiation to the lung that is >30 Gray (Gy) within 6 months of the first dose of study treatment.
* Participant has completed palliative radiotherapy within 7 days of the first dose of study treatment.
* Participant is ineligible if any of the following hepatic characteristics are present:
* Alanine aminotransferase (ALT) >2.5 times upper limit of normal (ULN) without liver metastases/tumor infiltration.
* ALT >5 times ULN with liver metastases/tumor infiltration.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per Investigator assessment)
* Participant has a corrected QT interval (QTc) >450 milliseconds (msec) (or QTc >480 msec for participants with bundle branch block).
* Participant has had major surgery within 3 weeks of the first dose of study treatment or has not adequately recovered from any AEs (Grade <=1) and/or complications from any major surgery. Surgical implantation of a port catheter is not exclusionary.
* Participant has an additional malignancy or a history of prior malignancy, with the exception of adequately treated basal or squamous skin cancer, cervical carcinoma in situ, or bladder carcinoma in situ without evidence of disease, or had a malignancy treated with curative intent and with no evidence of disease recurrence for 5 years since the initiation of that therapy.
* Participant has known active brain metastases and/or leptomeningeal metastases. Participants who have received prior therapy for their brain metastases and have radiographically stable central nervous system disease may participate, provided they are neurologically stable for at least 2 weeks before study entry and must be off corticosteroids within 3 days prior to the first dose of study treatment. Stable brain metastases by this definition should be established prior to the first dose of study treatment. Participants with known untreated, asymptomatic brain metastases (i.e., no neurological symptoms, no requirements for corticosteroids, no or minimal surrounding edema, and no lesions >1.5 centimeters [cm]) may participate, but will require regular imaging of the brain as a site of disease.
* Participant has tested positive for the presence of hepatitis B surface antigen or has a positive hepatitis C antibody test result at Screening, or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, participants who test positive for the presence of hepatitis B core antibody should also be excluded.
* Participant has an active infection requiring systemic therapy within 1 week prior to the anticipated first dose of study treatment.
* Participant has known human immunodeficiency virus (HIV) (positive for HIV 1 or HIV 2 antibodies).
* Participant has active autoimmune disease that required systemic treatment in the past 2 years, is immunocompromised in the opinion of the Investigator, or is receiving systemic immunosuppressive treatment. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Participant has received systemic steroid therapy within 3 days prior to the first dose of the study treatment or is receiving any other form of immunosuppressive medication. Replacement therapy is not considered a form of systemic therapy. Use of inhaled corticosteroids, local steroid injection, or steroid eye drops is allowed.
* Participant has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment of these conditions (including therapeutic thoraco or paracentesis) is eligible.
* Participant has current interstitial lung disease, current pneumonitis, or a history of pneumonitis that required the use of oral or IV glucocorticoids to assist with management. Lymphangitic spread of the NSCLC is not exclusionary.
* Participant has a history or current evidence of any medical condition, therapy, or laboratory abnormality that might confound the study results, interfere with their participation for the full duration of the study treatment, or indicate it is not in the best interest of the participant to participate, in the opinion of the Investigator.
* Participant has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, or peritoneal carcinomatosis.
* Participant has preexisting peripheral neuropathy that is Grade >=2 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 criteria.
* Participant has received a live vaccine within 30 days of the first dose of study treatment. Seasonal flu vaccines that do not contain live virus are permitted.
* Participant does not meet requirements per local prescribing guidelines for receiving treatment with either pemetrexed and cisplatin or carboplatin.
* Participant has sensitivity to any of the study treatments, or components thereof, or a history of drug or other allergy that, in the opinion of the Investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Participant is unable to interrupt aspirin or other nonsteroidal antiinflammatory drugs (NSAIDs), other than an aspirin dose <=1.3 gram (g) per day, for a 5 day period (8 day period for long acting agents, such as piroxicam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (3):
  - GSK Investigational Site, Denver, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Fairfax, Virginia
- Argentina (10):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Florida
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, La Rioja
  - GSK Investigational Site, Pergamino
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, Viedma
- Brazil (6):
  - GSK Investigational Site, Barretos
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, Natal
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- GSK Investigational Site, Santiago, Chile
- France (6):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Valenciennes
- Germany (5):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Immenhausen
  - GSK Investigational Site, Oldenburg
- Italy (5):
  - GSK Investigational Site, Aviano PN
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Roma
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
- South Korea (3):
  - GSK Investigational Site, Cheongju Chungcheongbuk-do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville
- Taiwan (2):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Austin D, Melhem M, Gandhi Y, Lu S, Visser S. Comparative analysis of PD-1 target engagement of dostarlimab and pembrolizumab in advanced solid tumors using ex vivo IL-2 stimulation data. CPT Pharmacometrics Syst Pharmacol. 2023 Jan;12(1):87-94. doi: 10.1002/psp4.12878. Epub 2022 Nov 16. PMID 36317409
- [Background] Lim SM, Peters S, Ortega Granados AL, Pinto GDJ, Fuentes CS, Lo Russo G, Schenker M, Ahn JS, Reck M, Szijgyarto Z, Huseinovic N, Zografos E, Buss E, Stjepanovic N, O'Donnell S, de Marinis F. Dostarlimab or pembrolizumab plus chemotherapy in previously untreated metastatic non-squamous non-small cell lung cancer: the randomized PERLA phase II trial. Nat Commun. 2023 Nov 11;14(1):7301. doi: 10.1038/s41467-023-42900-4. PMID 37951954
- [Derived] Lim SM, Ortega Granados AL, Pinto GDJ, Fuentes CS, Lo Russo G, Schenker M, Ahn JS, de Marinis F, Locke K Jr, Szijgyarto Z, Buss E, Stjepanovic N, Diaz-Padilla I, Peters S. Long-term Survival Analysis From PERLA, A Phase II Randomized Trial of Dostarlimab With Chemotherapy Versus Pembrolizumab With Chemotherapy in Metastatic Nonsquamous NSCLC. JTO Clin Res Rep. 2025 Sep 4;6(10):100900. doi: 10.1016/j.jtocrr.2025.100900. eCollection 2025 Oct. PMID 41080090

RESULTS

PARTICIPANT FLOW:
Groups:
- Dostarlimab + Chemotherapy: Participants with metastatic non-squamous non-small cell lung cancer (NSCLC) received dostarlimab and chemotherapy on Day 1 of every 21-day cycle beginning with Cycle 1. The order of administration of the investigational treatments was: dostarlimab first, immediately followed by pemetrexed, followed by cisplatin or carboplatin (Cycles 1 to 4 only). 500 milligram (mg) of dostarlimab was administered as a 30-minute intravenous (IV) infusion every three weeks (Q3W). 500 mg/meter^2 (m^2) pemetrexed was administered as a 10-minute IV infusion Q3W. 75 mg/m^2 cisplatin was administered via IV infusion approximately 30 minutes after pemetrexed infusion for Q3W or carboplatin at area under the concentration-time curve (AUC) 5 mg/milliliter/minute Q3W immediately following the pemetrexed infusion.
- Pembrolizumab + Chemotherapy: Participants with metastatic NSCLC received pembrolizumab and chemotherapy on Day 1 of every 21-day cycle beginning with Cycle 1. The order of administration of the investigational treatments was: pembrolizumab first, immediately followed by pemetrexed, followed by cisplatin or carboplatin (Cycles 1 to 4 only). 200 mg of pembrolizumab was administered as a 30-minute IV infusion Q3W. 500 mg/meter^2 (m^2) pemetrexed was administered as a 10-minute IV infusion Q3W. 75 mg/m^2 cisplatin was administered via IV infusion approximately 30 minutes after pemetrexed infusion for Q3W or carboplatin at area under the concentration-time curve (AUC) 5 mg/milliliter/minute Q3W immediately following the pemetrexed infusion.
Period: Overall Study
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Started | 121 | 122
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 81 (1 participant completed the follow-up and 80 participants died.) | 92 (1 participant completed the follow-up and 91 participants died.)
Not Completed | 40 | 30
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Study terminated by sponsor | 37 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy | Total
Number analyzed (Participants) | 121 | 122 | 243
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 63.4 (9.43) | 65.4 (8.51) | 64.4 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 45 | 81
  Male | 85 | 77 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 23 | 21 | 44
  Black or African American | 1 | 3 | 4
  White | 87 | 84 | 171
  Multiple | 3 | 3 | 6
  Not Reported | 2 | 5 | 7
  Unknown | 4 | 6 | 10

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death by any cause.
Time Frame: Up to approximately 46 months
Population: Intent-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Months | 20.2 [14.5 to 27.3] | 15.9 [11.6 to 19.3]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of disease progression (PD) or death by any cause, whichever occurs first. PFS was evaluated using Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1 based on Investigator assessment. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start).
Time Frame: Up to approximately 46 months
Population: Intent-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Months | 8.8 [6.9 to 11.0] | 6.8 [4.9 to 7.1]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAEs), TEAEs Leading to Death and TEAEs Leading to Treatment Discontinuation
Description: AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state. Number of participants with TEAEs, TEAEs leading to death, and TEAEs leading to treatment discontinuation are presented. AEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to 46 months
Population: Safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Participants
  TEAEs | 119 | 119
  TEAEs leading to death | 17 | 12
  TEAEs leading to treatment discontinuation | 35 | 46

4. Secondary Outcome: Number of Participants With Treatment Emergent Immune-related Adverse Event (irAE)
Description: The irAEs are events which are severe or fatal and can occur in participants treated with monoclonal antibodies directed against immune checkpoints, including pembrolizumab and dostarlimab. While irAEs (eg, diarrhea/colitis, pneumonitis, nephritis, hypophysitis, adrenalitis, thyroiditis, severe skin reactions, uveitis, myocarditis, and hepatotoxicity) usually occur during treatment, symptoms can also manifest after discontinuation of treatment. AEs were coded using the MedDRA dictionary.
Time Frame: Up to 46 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Participants | 38 | 47

5. Secondary Outcome: Number of Participants With Serious AEs
Description: An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the above outcomes. SAEs are subset of AEs. AEs were coded using the MedDRA dictionary.
Time Frame: Up to approximately 46 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Participants | 51 | 61

6. Secondary Outcome: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 30 to 110 units per liter (U/L) (Amylase); 4. 5 to 5. 6 milligram/deciliters (mg/dL) (Calcium); 96 to 100 milliequivalents (mEq)/ L (Chloride); 2. 5 to 4.5 mg/dL (Phosphate); 6 to 8.3 grams/L (protein); 6 to 24 millimoles/L (Urea) and 7 to 20 mg/dL (Urea nitrogen). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 117 | 115
Participants
  Amylase, To Low: number analyzed (Participants) | 116 | 114
  Amylase, To Low | 8 | 11
  Amylase, To Normal or No Change: number analyzed (Participants) | 116 | 114
  Amylase, To Normal or No Change | 76 | 76
  Amylase, To High: number analyzed (Participants) | 116 | 114
  Amylase, To High | 34 | 30
  Calcium, To Low | 42 | 39
  Calcium, To Normal or No Change | 60 | 65
  Calcium, To High | 25 | 16
  Chloride, To Low | 34 | 26
  Chloride, To Normal or No Change | 65 | 69
  Chloride, To High | 22 | 25
  Phosphate, To Low: number analyzed (Participants) | 117 | 114
  Phosphate, To Low | 32 | 22
  Phosphate, To Normal or No Change: number analyzed (Participants) | 117 | 114
  Phosphate, To Normal or No Change | 64 | 70
  Phosphate, To High: number analyzed (Participants) | 117 | 114
  Phosphate, To High | 26 | 28
  Protein, To Low: number analyzed (Participants) | 116 | 115
  Protein, To Low | 52 | 54
  Protein, To Normal or No Change: number analyzed (Participants) | 116 | 115
  Protein, To Normal or No Change | 55 | 56
  Protein, To High: number analyzed (Participants) | 116 | 115
  Protein, To High | 12 | 6
  Urea, To Low: number analyzed (Participants) | 89 | 90
  Urea, To Low | 7 | 11
  Urea, To Normal or No Change: number analyzed (Participants) | 89 | 90
  Urea, To Normal or No Change | 43 | 45
  Urea, To High: number analyzed (Participants) | 89 | 90
  Urea, To High | 41 | 37
  Urea Nitrogen, To Low: number analyzed (Participants) | 50 | 35
  Urea Nitrogen, To Low | 5 | 6
  Urea Nitrogen, To Normal or No Change: number analyzed (Participants) | 50 | 35
  Urea Nitrogen, To Normal or No Change | 26 | 17
  Urea Nitrogen, To High: number analyzed (Participants) | 50 | 35
  Urea Nitrogen, To High | 20 | 13

7. Secondary Outcome: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.01 to 0.3*10^9 cells/L (basophils); 41 to 50 percentage of red blood cells (RBC) in blood (hematocrit); 80-100 femtoliters (fl) (erythrocytes [referred as Ery] mean corpuscular volume (EMCV)); 2 to 8 percentage of WBC (monocytes); and Women: 4.2 to 5.4 million RBC/ microliter (mcL) of blood and Men: 4.7 to 6.1 million RBC/ mcL (erythrocytes). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 118 | 115
Participants
  Basophils, To Low: number analyzed (Participants) | 101 | 102
  Basophils, To Low | 12 | 9
  Basophils, To Normal or No Change: number analyzed (Participants) | 101 | 102
  Basophils, To Normal or No Change | 72 | 75
  Basophils, To High: number analyzed (Participants) | 101 | 102
  Basophils, To High | 19 | 19
  Hematocrit, To Low | 73 | 64
  Hematocrit, To Normal or No Change | 43 | 50
  Hematocrit, To High | 3 | 1
  EMCV, To Low | 6 | 11
  EMCV, To Normal or No Change | 59 | 54
  EMCV, To High | 57 | 54
  Monocytes, To Low: number analyzed (Participants) | 101 | 102
  Monocytes, To Low | 23 | 21
  Monocytes, To Normal or No Change: number analyzed (Participants) | 101 | 102
  Monocytes, To Normal or No Change | 41 | 42
  Monocytes, To High: number analyzed (Participants) | 101 | 102
  Monocytes, To High | 46 | 43
  Erythrocytes, To Low | 73 | 79
  Erythrocytes, To Normal or No Change | 44 | 34
  Erythrocytes, To High | 2 | 6

8. Secondary Outcome: Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline
Description: Urine samples were collected to assess urine Bilirubin, glucose, ketones, Leukocyte Esterase, Nitrite, occult blood and Protein using dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as No Change/Decreased, Increase to TRACE, Increase to +, Increase to ++, Increase to +++ and Increase to ++++. Baseline (Day 1) was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 93 | 71
Participants
  Bilirubin, No Change/Decreased: number analyzed (Participants) | 90 | 69
  Bilirubin, No Change/Decreased | 86 | 66
  Bilirubin, Increase to TRACE: number analyzed (Participants) | 90 | 69
  Bilirubin, Increase to TRACE | 0 | 0
  Bilirubin, Increase to +: number analyzed (Participants) | 90 | 69
  Bilirubin, Increase to + | 4 | 3
  Bilirubin, Increase to ++: number analyzed (Participants) | 90 | 69
  Bilirubin, Increase to ++ | 0 | 0
  Bilirubin, Increase to +++: number analyzed (Participants) | 90 | 69
  Bilirubin, Increase to +++ | 0 | 0
  Bilirubin, Increase to ++++: number analyzed (Participants) | 90 | 69
  Bilirubin, Increase to ++++ | 0 | 0
  Glucose, No Change/Decreased | 79 | 57
  Glucose, Increase to TRACE | 2 | 1
  Glucose, Increase to + | 8 | 8
  Glucose, Increase to ++ | 1 | 2
  Glucose, Increase to +++ | 1 | 2
  Glucose, Increase to ++++ | 2 | 1
  Ketones, No Change/Decreased | 81 | 58
  Ketones, Increase to TRACE | 4 | 3
  Ketones, Increase to + | 8 | 7
  Ketones, Increase to ++ | 0 | 2
  Ketones, Increase to +++ | 0 | 1
  Ketones, Increase to ++++ | 0 | 0
  Leukocyte Esterase, No Change/Decreased: number analyzed (Participants) | 91 | 70
  Leukocyte Esterase, No Change/Decreased | 75 | 55
  Leukocyte Esterase, Increase to TRACE: number analyzed (Participants) | 91 | 70
  Leukocyte Esterase, Increase to TRACE | 1 | 2
  Leukocyte Esterase, Increase to +: number analyzed (Participants) | 91 | 70
  Leukocyte Esterase, Increase to + | 11 | 10
  Leukocyte Esterase, Increase to ++: number analyzed (Participants) | 91 | 70
  Leukocyte Esterase, Increase to ++ | 2 | 0
  Leukocyte Esterase, Increase to +++: number analyzed (Participants) | 91 | 70
  Leukocyte Esterase, Increase to +++ | 1 | 3
  Leukocyte Esterase, Increase to ++++: number analyzed (Participants) | 91 | 70
  Leukocyte Esterase, Increase to ++++ | 1 | 0
  Nitrite, No Change/Decreased | 90 | 70
  Nitrite, Increase to TRACE | 0 | 0
  Nitrite, Increase to + | 3 | 1
  Nitrite, Increase to ++ | 0 | 0
  Nitrite, Increase to +++ | 0 | 0
  Nitrite, Increase to ++++ | 0 | 0
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 92 | 71
  Occult Blood, No Change/Decreased | 77 | 57
  Occult Blood, Increase to TRACE: number analyzed (Participants) | 92 | 71
  Occult Blood, Increase to TRACE | 6 | 3
  Occult Blood, Increase to +: number analyzed (Participants) | 92 | 71
  Occult Blood, Increase to + | 6 | 8
  Occult Blood, Increase to ++: number analyzed (Participants) | 92 | 71
  Occult Blood, Increase to ++ | 3 | 3
  Occult Blood, Increase to +++: number analyzed (Participants) | 92 | 71
  Occult Blood, Increase to +++ | 0 | 0
  Occult Blood, Increase to ++++: number analyzed (Participants) | 92 | 71
  Occult Blood, Increase to ++++ | 0 | 0
  Protein, No Change/Decreased: number analyzed (Participants) | 93 | 70
  Protein, No Change/Decreased | 71 | 53
  Protein, Increase to TRACE: number analyzed (Participants) | 93 | 70
  Protein, Increase to TRACE | 7 | 3
  Protein, Increase to +: number analyzed (Participants) | 93 | 70
  Protein, Increase to + | 14 | 10
  Protein, Increase to ++: number analyzed (Participants) | 93 | 70
  Protein, Increase to ++ | 0 | 3
  Protein, Increase to +++: number analyzed (Participants) | 93 | 70
  Protein, Increase to +++ | 1 | 1
  Protein, Increase to ++++: number analyzed (Participants) | 93 | 70
  Protein, Increase to ++++ | 0 | 0

9. Secondary Outcome: Change From Baseline (CFB) in Thyroid Functions: Free Triiodothyronine (T3) and Free Thyroxine (T4)
Description: Blood samples were collected for the assessment Free Triiodothyronine (T3) and Free Thyroxine (T4).
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed
Measure: Mean (Standard Deviation); unit: Picomoles per liter(pmol/L)
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 90 | 106
Picomoles per liter(pmol/L)
  Triiodothyronine, Free, Baseline: number analyzed (Participants) | 79 | 91
  Triiodothyronine, Free, Baseline | 4.48026 (1.638746) | 4.48540 (1.066597)
  Triiodothyronine, Free, CFB to Cycle 2 Day 1: number analyzed (Participants) | 55 | 63
  Triiodothyronine, Free, CFB to Cycle 2 Day 1 | -0.12423 (2.071042) | -0.24330 (1.026993)
  Triiodothyronine, Free, CFB to Cycle 4 Day 1: number analyzed (Participants) | 48 | 54
  Triiodothyronine, Free, CFB to Cycle 4 Day 1 | -0.00187 (2.206972) | -0.11796 (1.413190)
  Triiodothyronine, Free, CFB to Cycle 6 Day 1: number analyzed (Participants) | 50 | 48
  Triiodothyronine, Free, CFB to Cycle 6 Day 1 | -0.15030 (2.128584) | -0.37705 (1.117516)
  Triiodothyronine, Free, CFB to Cycle 8 Day 1: number analyzed (Participants) | 41 | 39
  Triiodothyronine, Free, CFB to Cycle 8 Day 1 | 0.11483 (2.738875) | -0.43073 (1.123017)
  Triiodothyronine, Free, CFB to Cycle 10 Day 1: number analyzed (Participants) | 44 | 31
  Triiodothyronine, Free, CFB to Cycle 10 Day 1 | -0.25993 (2.187046) | -0.23819 (1.273369)
  Triiodothyronine, Free, CFB to Cycle 12 Day 1: number analyzed (Participants) | 38 | 30
  Triiodothyronine, Free, CFB to Cycle 12 Day 1 | -0.04347 (2.817465) | 5.82171 (34.328615)
  Triiodothyronine, Free, CFB to Cycle 14 Day 1: number analyzed (Participants) | 30 | 25
  Triiodothyronine, Free, CFB to Cycle 14 Day 1 | -0.61895 (2.558169) | -0.33501 (1.597219)
  Triiodothyronine, Free, CFB to Cycle 16 Day 1: number analyzed (Participants) | 27 | 28
  Triiodothyronine, Free, CFB to Cycle 16 Day 1 | -0.44645 (2.274173) | -0.36614 (1.108135)
  Triiodothyronine, Free, CFB to Cycle 18 Day 1: number analyzed (Participants) | 24 | 20
  Triiodothyronine, Free, CFB to Cycle 18 Day 1 | -0.37234 (2.414983) | -0.12607 (1.337185)
  Triiodothyronine, Free, CFB to Cycle 20 Day 1: number analyzed (Participants) | 25 | 18
  Triiodothyronine, Free, CFB to Cycle 20 Day 1 | -0.37506 (2.495642) | -0.26936 (1.237097)
  Triiodothyronine, Free, CFB to Cycle 22 Day 1: number analyzed (Participants) | 22 | 21
  Triiodothyronine, Free, CFB to Cycle 22 Day 1 | -0.36400 (2.759103) | -0.17980 (1.018812)
  Triiodothyronine, Free, CFB to Cycle 24 Day 1: number analyzed (Participants) | 20 | 19
  Triiodothyronine, Free, CFB to Cycle 24 Day 1 | -0.69144 (2.662922) | -0.18380 (0.736262)
  Triiodothyronine, Free, CFB to Cycle 26 Day 1: number analyzed (Participants) | 19 | 18
  Triiodothyronine, Free, CFB to Cycle 26 Day 1 | 0.01392 (1.331466) | -0.39401 (0.669173)
  Triiodothyronine, Free, CFB to Cycle 28 Day 1: number analyzed (Participants) | 19 | 15
  Triiodothyronine, Free, CFB to Cycle 28 Day 1 | -0.05502 (1.094085) | -0.28233 (0.880805)
  Triiodothyronine, Free, CFB to Cycle 30 Day 1: number analyzed (Participants) | 18 | 15
  Triiodothyronine, Free, CFB to Cycle 30 Day 1 | 0.11929 (1.151771) | -0.19119 (0.911551)
  Triiodothyronine, Free, CFB to Cycle 32 Day 1: number analyzed (Participants) | 16 | 14
  Triiodothyronine, Free, CFB to Cycle 32 Day 1 | 0.54114 (1.043916) | 0.03556 (1.067239)
  Triiodothyronine, Free, CFB to Cycle 34 Day 1: number analyzed (Participants) | 13 | 11
  Triiodothyronine, Free, CFB to Cycle 34 Day 1 | 0.62534 (0.957105) | -0.32236 (0.774334)
  Triiodothyronine, Free, CFB to End of Treatment: number analyzed (Participants) | 48 | 48
  Triiodothyronine, Free, CFB to End of Treatment | -0.64275 (2.184114) | -0.40528 (1.086922)
  Thyroxine, Free, Baseline | 16.33405 (4.294246) | 15.93013 (3.436512)
  Thyroxine, Free, CFB to Cycle 2 Day 1: number analyzed (Participants) | 68 | 72
  Thyroxine, Free, CFB to Cycle 2 Day 1 | -0.35227 (4.257866) | 0.21349 (3.541952)
  Thyroxine, Free, CFB to Cycle 4 Day 1: number analyzed (Participants) | 60 | 65
  Thyroxine, Free, CFB to Cycle 4 Day 1 | 0.04265 (6.245167) | 0.08969 (4.015042)
  Thyroxine, Free, CFB to Cycle 6 Day 1: number analyzed (Participants) | 62 | 58
  Thyroxine, Free, CFB to Cycle 6 Day 1 | -0.10229 (5.418010) | -0.58695 (3.404576)
  Thyroxine, Free, CFB to Cycle 8 Day 1: number analyzed (Participants) | 52 | 52
  Thyroxine, Free, CFB to Cycle 8 Day 1 | -1.02504 (6.168755) | 0.27944 (3.877876)
  Thyroxine, Free, CFB to Cycle 10 Day 1: number analyzed (Participants) | 52 | 39
  Thyroxine, Free, CFB to Cycle 10 Day 1 | -1.15108 (5.586383) | 0.08349 (3.613602)
  Thyroxine, Free, CFB to Cycle 12 Day 1: number analyzed (Participants) | 47 | 35
  Thyroxine, Free, CFB to Cycle 12 Day 1 | -0.16670 (6.081753) | 4.71828 (27.489015)
  Thyroxine, Free, CFB to Cycle 14 Day 1: number analyzed (Participants) | 35 | 32
  Thyroxine, Free, CFB to Cycle 14 Day 1 | 0.32703 (6.114475) | -0.45213 (4.196576)
  Thyroxine, Free, CFB to Cycle 16 Day 1: number analyzed (Participants) | 31 | 34
  Thyroxine, Free, CFB to Cycle 16 Day 1 | -0.45337 (4.840440) | 0.24537 (3.472618)
  Thyroxine, Free, CFB to Cycle 18 Day 1: number analyzed (Participants) | 31 | 25
  Thyroxine, Free, CFB to Cycle 18 Day 1 | 0.07645 (5.524789) | 0.47690 (1.984139)
  Thyroxine, Free, CFB to Cycle 20 Day 1: number analyzed (Participants) | 31 | 24
  Thyroxine, Free, CFB to Cycle 20 Day 1 | -0.41084 (5.013270) | 0.37830 (3.413511)
  Thyroxine, Free, CFB to Cycle 22 Day 1: number analyzed (Participants) | 27 | 25
  Thyroxine, Free, CFB to Cycle 22 Day 1 | -0.65956 (5.562802) | 0.45462 (2.841910)
  Thyroxine, Free, CFB to Cycle 24 Day 1: number analyzed (Participants) | 24 | 22
  Thyroxine, Free, CFB to Cycle 24 Day 1 | -0.71092 (6.314352) | 0.31032 (2.653193)
  Thyroxine, Free, CFB to Cycle 26 Day 1: number analyzed (Participants) | 22 | 22
  Thyroxine, Free, CFB to Cycle 26 Day 1 | -0.89968 (5.246300) | 0.23139 (3.443957)
  Thyroxine, Free, CFB to Cycle 28 Day 1: number analyzed (Participants) | 22 | 20
  Thyroxine, Free, CFB to Cycle 28 Day 1 | -0.89658 (5.489130) | 1.10907 (2.849631)
  Thyroxine, Free, CFB to Cycle 30 Day 1: number analyzed (Participants) | 20 | 18
  Thyroxine, Free, CFB to Cycle 30 Day 1 | -1.46126 (4.811596) | -0.21286 (3.203649)
  Thyroxine, Free, CFB to Cycle 32 Day 1: number analyzed (Participants) | 18 | 16
  Thyroxine, Free, CFB to Cycle 32 Day 1 | -1.81377 (5.474197) | 0.13236 (3.519557)
  Thyroxine, Free, CFB to Cycle 34 Day 1: number analyzed (Participants) | 16 | 15
  Thyroxine, Free, CFB to Cycle 34 Day 1 | -1.52641 (6.379163) | 0.45041 (2.435328)
  Thyroxine, Free, CFB to End of Treatment: number analyzed (Participants) | 58 | 62
  Thyroxine, Free, CFB to End of Treatment | 0.26660 (3.882315) | 0.46964 (3.310829)

10. Secondary Outcome: Change From Baseline in Thyroid Function: Thyrotropin (TSH)
Description: Blood samples were collected for the assessment of Thyroid Function Thyrotropin (TSH).
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed
Measure: Mean (Standard Deviation); unit: Milli-international Units/ Liter
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 116 | 120
Milli-international Units/ Liter
  Baseline | 1.853 (1.8354) | 1.904 (1.7421)
  CFB to Cycle 2 Day 1: number analyzed (Participants) | 93 | 87
  CFB to Cycle 2 Day 1 | 0.225 (3.7642) | -0.497 (1.7405)
  CFB to Cycle 4 Day 1: number analyzed (Participants) | 87 | 79
  CFB to Cycle 4 Day 1 | 1.285 (9.4283) | -0.622 (1.7892)
  CFB to Cycle 6 Day 1: number analyzed (Participants) | 85 | 66
  CFB to Cycle 6 Day 1 | 1.123 (8.4596) | 2.006 (21.0213)
  CFB to Cycle 8 Day 1: number analyzed (Participants) | 68 | 61
  CFB to Cycle 8 Day 1 | 2.454 (9.7235) | 2.648 (22.9952)
  CFB to Cycle 10 Day 1: number analyzed (Participants) | 67 | 49
  CFB to Cycle 10 Day 1 | 3.233 (12.1571) | 1.986 (12.8377)
  CFB to Cycle 12 Day 1: number analyzed (Participants) | 63 | 43
  CFB to Cycle 12 Day 1 | 2.448 (9.8590) | 1.138 (10.9780)
  CFB to Cycle 14 Day 1: number analyzed (Participants) | 49 | 39
  CFB to Cycle 14 Day 1 | 1.282 (4.2566) | 1.734 (9.0539)
  CFB to Cycle 16 Day 1: number analyzed (Participants) | 47 | 39
  CFB to Cycle 16 Day 1 | 1.551 (4.7982) | 2.056 (13.4532)
  CFB to Cycle 18 Day 1: number analyzed (Participants) | 43 | 30
  CFB to Cycle 18 Day 1 | 1.190 (4.1837) | -0.406 (1.6364)
  CFB to Cycle 20 Day 1: number analyzed (Participants) | 42 | 29
  CFB to Cycle 20 Day 1 | 1.685 (5.3517) | 1.825 (11.8029)
  CFB to Cycle 22 Day 1: number analyzed (Participants) | 38 | 29
  CFB to Cycle 22 Day 1 | 1.428 (5.9512) | 1.794 (10.5658)
  CFB to Cycle 24 Day 1: number analyzed (Participants) | 34 | 25
  CFB to Cycle 24 Day 1 | 0.993 (3.0372) | 2.161 (10.7015)
  CFB to Cycle 26 Day 1: number analyzed (Participants) | 28 | 25
  CFB to Cycle 26 Day 1 | 1.029 (4.3080) | 2.050 (11.8067)
  CFB to Cycle 28 Day 1: number analyzed (Participants) | 29 | 23
  CFB to Cycle 28 Day 1 | 1.204 (3.4902) | 1.760 (9.6622)
  CFB to Cycle 30 Day 1: number analyzed (Participants) | 26 | 21
  CFB to Cycle 30 Day 1 | 1.615 (5.4966) | 3.468 (15.7231)
  CFB to Cycle 32 Day 1: number analyzed (Participants) | 23 | 17
  CFB to Cycle 32 Day 1 | 1.824 (4.9423) | 0.365 (0.8151)
  CFB to Cycle 34 Day 1: number analyzed (Participants) | 20 | 17
  CFB to Cycle 34 Day 1 | 1.081 (2.4504) | -0.189 (1.5062)
  CFB to End of Treatment: number analyzed (Participants) | 75 | 77
  CFB to End of Treatment | 2.210 (8.3867) | 1.303 (9.3590)

11. Secondary Outcome: Change From Baseline in Thyroid Functions: Triiodothyronine (T3) and Thyroxine (T4)
Description: Blood samples were collected for the assessment of Triiodothyronine (T3) and Thyroxine (T4).
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed
Measure: Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 27 | 22
Nanomoles per liter (nmol/L)
  Triiodothyronine, Baseline: number analyzed (Participants) | 9 | 6
  Triiodothyronine, Baseline | 1.68399 (0.308404) | 1.48287 (0.526037)
  Triiodothyronine, CFB to Cycle 2 Day 1: number analyzed (Participants) | 4 | 1
  Triiodothyronine, CFB to Cycle 2 Day 1 | 0.06903 (0.172873) | -0.58292
  Triiodothyronine, CFB to Cycle 4 Day 1: number analyzed (Participants) | 2 | 0
  Triiodothyronine, CFB to Cycle 4 Day 1 | -0.41878 (0.353613) |
  Triiodothyronine, CFB to Cycle 6 Day 1: number analyzed (Participants) | 1 | 0
  Triiodothyronine, CFB to Cycle 6 Day 1 | -0.21476 |
  Thyroxine, Baseline | 72.72912 (46.845564) | 85.29069 (38.027652)
  Thyroxine, CFB to Cycle 2 Day 1: number analyzed (Participants) | 23 | 14
  Thyroxine, CFB to Cycle 2 Day 1 | 16.06393 (38.489073) | -3.12689 (11.544100)
  Thyroxine, CFB to Cycle 4 Day 1: number analyzed (Participants) | 24 | 12
  Thyroxine, CFB to Cycle 4 Day 1 | 10.16002 (47.746764) | 12.22592 (30.578995)
  Thyroxine, CFB to Cycle 6 Day 1: number analyzed (Participants) | 19 | 10
  Thyroxine, CFB to Cycle 6 Day 1 | 9.83083 (30.658114) | -2.45916 (27.497527)
  Thyroxine, CFB to Cycle 8 Day 1: number analyzed (Participants) | 15 | 9
  Thyroxine, CFB to Cycle 8 Day 1 | 21.85010 (44.242770) | -0.06812 (24.146111)
  Thyroxine, CFB to Cycle 10 Day 1: number analyzed (Participants) | 14 | 8
  Thyroxine, CFB to Cycle 10 Day 1 | 32.19186 (41.441071) | -0.03002 (16.413851)
  Thyroxine, CFB to Cycle 12 Day 1: number analyzed (Participants) | 13 | 6
  Thyroxine, CFB to Cycle 12 Day 1 | 23.45510 (36.165686) | -0.82919 (9.539787)
  Thyroxine, CFB to Cycle 14 Day 1: number analyzed (Participants) | 11 | 6
  Thyroxine, CFB to Cycle 14 Day 1 | 14.79794 (35.614508) | 0.64908 (12.623292)
  Thyroxine, CFB to Cycle 16 Day 1: number analyzed (Participants) | 8 | 4
  Thyroxine, CFB to Cycle 16 Day 1 | 21.23230 (38.220665) | 7.86174 (18.910608)
  Thyroxine, CFB to Cycle 18 Day 1: number analyzed (Participants) | 7 | 4
  Thyroxine, CFB to Cycle 18 Day 1 | 18.35801 (31.436316) | 7.37470 (8.635752)
  Thyroxine, CFB to Cycle 20 Day 1: number analyzed (Participants) | 6 | 4
  Thyroxine, CFB to Cycle 20 Day 1 | 26.94600 (47.915257) | 16.06215 (18.656008)
  Thyroxine, CFB to Cycle 22 Day 1: number analyzed (Participants) | 7 | 4
  Thyroxine, CFB to Cycle 22 Day 1 | 22.73866 (34.202890) | 18.57057 (22.383758)
  Thyroxine, CFB to Cycle 24 Day 1: number analyzed (Participants) | 6 | 3
  Thyroxine, CFB to Cycle 24 Day 1 | 24.31027 (45.963345) | 23.08569 (20.160509)
  Thyroxine, CFB to Cycle 26 Day 1: number analyzed (Participants) | 4 | 2
  Thyroxine, CFB to Cycle 26 Day 1 | 32.22436 (62.122105) | 35.71425 (12.285627)
  Thyroxine, CFB to Cycle 28 Day 1: number analyzed (Participants) | 6 | 3
  Thyroxine, CFB to Cycle 28 Day 1 | 21.13316 (46.351292) | 20.55189 (17.985775)
  Thyroxine, CFB to Cycle 30 Day 1: number analyzed (Participants) | 5 | 3
  Thyroxine, CFB to Cycle 30 Day 1 | 19.12904 (53.351526) | 13.09008 (11.862148)
  Thyroxine, CFB to Cycle 32 Day 1: number analyzed (Participants) | 4 | 2
  Thyroxine, CFB to Cycle 32 Day 1 | 19.99271 (58.500079) | 16.73184 (23.660023)
  Thyroxine, CFB to Cycle 34 Day 1: number analyzed (Participants) | 3 | 1
  Thyroxine, CFB to Cycle 34 Day 1 | -4.97280 (8.622499) | 0.01300
  Thyroxine, CFB to End of Treatment: number analyzed (Participants) | 14 | 10
  Thyroxine, CFB to End of Treatment | 11.06954 (35.792455) | 4.67311 (29.791225)

12. Secondary Outcome: Number of Participants With Worst-case Grade Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in a semi-supine position after 5 minutes rest. Grades were derived based on numeric criteria as defined in Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Systolic Blood Pressure (SBP): Grade 0 (<120 Millimetre of mercury (mmHg)), Grade 1 (120-139 mmHg), Grade 2 (140-159 mmHg), Grade 3 (>=160 mmHg). Diastolic Blood Pressure (DBP): Grade 0 (<80 mmHg), Grade 1 (80-89 mmHg), Grade 2 (90-99 mmHg), Grade 3 (>=100 mmHg). An increase is defined as an increase in the CTCAE grade relative to the Baseline grade. Only those participants with grade increase have been presented. Participants with missing Baseline values were assumed to have a Baseline value of G0.
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 117 | 115
Participants
  DBP, Increase to Grade 1 | 36 | 27
  DBP, Increase to Grade 2 | 35 | 25
  DBP, Increase to Grade 3 | 6 | 7
  SBP, Increase to Grade 1 | 24 | 18
  SBP, Increase to Grade 2 | 34 | 24
  SBP, Increase to Grade 3 | 8 | 11

13. Secondary Outcome: Number of Participants With Worst Case Pulse Rate Results Post-Baseline Relative to Baseline Based on Potential Clinical Importance (PCI)
Description: Normal range of Pulse Rate was 60 to 100 beats/min. Participants were counted in worst case category that their value changes to low, to within [w/in] Range or No Change [NC] or high, unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category.
Time Frame: Up to approximately 46 months
Population: Safety population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 117 | 115
Participants
  To Low | 5 | 3
  To w/in Range or No Change | 105 | 103
  To High | 7 | 9

14. Secondary Outcome: Number of Participants With Worst-Case Post-Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Performance status was assessed using the ECOG scale (Grade 0-5). Grades: 0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory, able to carry out work of light nature. 2: Ambulatory, capable of self-care, unable to carry out work activities. Up and about more than 50% waking hours. 3: Capable of limited self-care, confined to bed/chair more than 50% waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair. 5: Dead.
Time Frame: Up to approximately 46 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 118 | 115
Participants
  0 | 15 | 20
  1 | 70 | 57
  2 | 24 | 20
  3 | 4 | 14
  4-5 | 5 | 4

15. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters
Description: Participants were in a supine or semi recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs were recorded. Single 12-lead ECG was recorded using an ECG machine. PR, QRS, QT, QTcF, and RR intervals were recorded
Time Frame: Baseline (Day 1), Cycle 1 Day 1, and end of treatment (Up to approximately 46 months)
Population: Safety population. Only those participants with data available at specified categories have been analyzed
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Millisecond (msec)
  PR Interval, Baseline: number analyzed (Participants) | 120 | 119
  PR Interval, Baseline | 157.3 (26.87) | 152.4 (25.54)
  PR Interval, CFB to Cycle 1 Day 1: number analyzed (Participants) | 2 | 3
  PR Interval, CFB to Cycle 1 Day 1 | -6.0 (1.41) | 8.7 (16.17)
  PR Interval, CFB to End of Treatment: number analyzed (Participants) | 79 | 67
  PR Interval, CFB to End of Treatment | -5.3 (23.35) | 0.2 (17.49)
  QRS Duration, Baseline | 87.9 (14.85) | 89.0 (14.91)
  QRS Duration, CFB to Cycle 1 Day 1: number analyzed (Participants) | 3 | 2
  QRS Duration, CFB to Cycle 1 Day 1 | 10.0 (13.08) | 6.0 (14.14)
  QRS Duration, CFB to End of Treatment: number analyzed (Participants) | 79 | 69
  QRS Duration, CFB to End of Treatment | 3.3 (17.14) | -1.1 (13.47)
  QT Interval, Baseline | 370.4 (35.29) | 374.3 (38.05)
  QT Interval, CFB to Cycle 1 Day 1: number analyzed (Participants) | 4 | 3
  QT Interval, CFB to Cycle 1 Day 1 | -19.5 (48.23) | -27.3 (57.98)
  QT Interval, CFB to End of Treatment: number analyzed (Participants) | 79 | 69
  QT Interval, CFB to End of Treatment | -1.7 (36.57) | -4.1 (38.07)
  QTcB Interval, Baseline: number analyzed (Participants) | 120 | 122
  QTcB Interval, Baseline | 459.3 (190.83) | 440.4 (121.20)
  QTcB Interval, CFB to Cycle 1 Day 1: number analyzed (Participants) | 3 | 3
  QTcB Interval, CFB to Cycle 1 Day 1 | -309.0 (559.52) | -31.7 (49.81)
  QTcB Interval, CFB to End of Treatment: number analyzed (Participants) | 77 | 70
  QTcB Interval, CFB to End of Treatment | -12.2 (176.21) | -3.1 (30.81)
  QTcF Interval, Baseline: number analyzed (Participants) | 119 | 121
  QTcF Interval, Baseline | 406.6 (50.60) | 412.9 (48.99)
  QTcF Interval, CFB to Cycle 1 Day 1: number analyzed (Participants) | 3 | 3
  QTcF Interval, CFB to Cycle 1 Day 1 | -12.3 (48.19) | -4.7 (4.16)
  QTcF Interval, CFB to End of Treatment: number analyzed (Participants) | 75 | 68
  QTcF Interval, CFB to End of Treatment | 1.4 (65.82) | -10.0 (60.00)
  RR Interval, Baseline: number analyzed (Participants) | 119 | 121
  RR Interval, Baseline | 741.3 (205.25) | 766.5 (195.43)
  RR Interval, CFB to Cycle 1 Day 1: number analyzed (Participants) | 3 | 3
  RR Interval, CFB to Cycle 1 Day 1 | 81.3 (256.20) | -10.7 (81.05)
  RR Interval, CFB to End of Treatment: number analyzed (Participants) | 75 | 68
  RR Interval, CFB to End of Treatment | -3.3 (183.71) | 2.5 (193.04)

16. Secondary Outcome: Mean Change From Baseline in ECG Mean Heart Rate
Description: Participants were in a supine or semi recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs were recorded. Single 12-lead ECG was recorded using an ECG machine. Mean Heart rate were recorded.
Time Frame: Baseline (Day 1), Cycle 1 Day 1, and end of treatment (Up to approximately 46 months)
Population: Safety population. Only those participants with data available at specified categories have been analyzed
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
beats/min
  Baseline | 79.8 (15.17) | 80.0 (16.14)
  CFB to Cycle 1 Day 1: number analyzed (Participants) | 4 | 3
  CFB to Cycle 1 Day 1 | 0.0 (13.04) | 3.3 (13.65)
  CFB to End of Treatment: number analyzed (Participants) | 79 | 70
  CFB to End of Treatment | 1.5 (14.71) | 0.6 (17.95)

17. Secondary Outcome: Number Participant Who Used Concomitant Medications
Description: Number of participants received concomitant medications were summarized.
Time Frame: Up to approximately 46 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Participants | 121 | 122

18. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or confirmed partial response (PR) as their best overall response (BOR) recorded from the date of randomization until disease progression or initiation of new anti-cancer therapy, whichever is earlier based on blinded independent central review (BICR) evaluation criteria in solid tumors (RECIST) version 1.1 (v1.1). CR was defined as disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters (e.g., percent change from baseline).
Time Frame: Up to approximately 20 months
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
Number analyzed (Participants) | 121 | 122
Percentage of Participants | 46 [37.2 to 55.6] | 37 [28.3 to 46.1]
Statistical Analysis 1: Comparison: Dostarlimab + Chemotherapy vs Pembrolizumab + Chemotherapy; Test type: Other; Difference in Response Rate = 9.32, 80% CI 2-sided [1.46 to 17.18] — Mantel and Haenszel method with Sato's variance estimator was used for between arms comparison and was stratified by PD-L1 status and smoking status based on the strata data collected in interactive response technology (IRT) at randomization

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from Day 1 and up to approximately 46 months.
Description: Safety population included all participants who received at least 1 dose of study treatment.
Arm/Group | Dostarlimab + Chemotherapy | Pembrolizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 80/121 | 91/122
Serious Adverse Events (participants affected / at risk) | 51/121 | 61/122
Other Adverse Events (participants affected / at risk) | 117/121 | 114/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dostarlimab + Chemotherapy (N=121) | Pembrolizumab + Chemotherapy (N=122)
Anaemia (Blood and lymphatic system disorders) | 9 (11) | 6 (7)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 3 (3) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (5) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 15 (15)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 2 (2)
Strongyloidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dostarlimab + Chemotherapy (N=121) | Pembrolizumab + Chemotherapy (N=122)
Anaemia (Blood and lymphatic system disorders) | 63 (194) | 59 (156)
Neutropenia (Blood and lymphatic system disorders) | 22 (42) | 25 (45)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (30) | 10 (15)
Hyperthyroidism (Endocrine disorders) | 8 (11) | 2 (3)
Hypothyroidism (Endocrine disorders) | 11 (13) | 7 (8)
Constipation (Gastrointestinal disorders) | 24 (37) | 26 (31)
Diarrhoea (Gastrointestinal disorders) | 21 (31) | 17 (20)
Nausea (Gastrointestinal disorders) | 31 (105) | 32 (66)
Stomatitis (Gastrointestinal disorders) | 8 (10) | 5 (5)
Vomiting (Gastrointestinal disorders) | 25 (38) | 16 (21)
Asthenia (General disorders) | 41 (99) | 42 (90)
Chest pain (General disorders) | 3 (3) | 8 (9)
Fatigue (General disorders) | 15 (37) | 16 (22)
Mucosal inflammation (General disorders) | 7 (9) | 7 (10)
Oedema peripheral (General disorders) | 14 (20) | 11 (22)
Pain (General disorders) | 7 (8) | 3 (3)
Pyrexia (General disorders) | 14 (21) | 15 (27)
COVID-19 (Infections and infestations) | 7 (7) | 9 (9)
Conjunctivitis (Infections and infestations) | 8 (14) | 6 (6)
Pneumonia (Infections and infestations) | 7 (11) | 8 (10)
Respiratory tract infection (Infections and infestations) | 7 (9) | 13 (16)
Alanine aminotransferase increased (Investigations) | 15 (26) | 14 (26)
Amylase increased (Investigations) | 6 (25) | 7 (13)
Aspartate aminotransferase increased (Investigations) | 12 (22) | 9 (19)
Blood alkaline phosphatase increased (Investigations) | 8 (11) | 8 (12)
Blood creatinine increased (Investigations) | 18 (22) | 9 (26)
Gamma-glutamyltransferase increased (Investigations) | 8 (14) | 6 (10)
Platelet count decreased (Investigations) | 2 (2) | 9 (21)
Weight decreased (Investigations) | 9 (11) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 24 (38) | 20 (22)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8) | 8 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (16) | 9 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (11) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (16) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 15 (18)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4)
Dizziness (Nervous system disorders) | 9 (11) | 6 (7)
Headache (Nervous system disorders) | 8 (13) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (33) | 22 (34)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (41) | 21 (33)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (19) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 16 (17) | 7 (8)
Hypertension (Vascular disorders) | 9 (20) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT04581824/Prot_004.pdf
  • Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04581824/SAP_005.pdf